CLINICAL TRIAL: NCT01986309
Title: Use of Intravenous Lidocaine in the Prevention of Postoperative Vomiting in Elective Tonsil Surgery, With or Without Adenoids
Brief Title: Intravenous Lidocaine in the Prevention of Postoperative Vomiting in Elective Tonsil Surgery
Acronym: LETSVN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PG 08-12
Record Dates: First submitted 2013-07-08; First posted 2013-11-18 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Postoperative Nausea and Vomiting; Pain
Keywords: Postoperative; Nausea; Vomiting; Pain; Surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain; Nausea; Vomiting | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group L (Active Comparator): Group L Lidocaine load dose 1.5 mg / kg over 5 minutes, followed by continuous infusion of 2 mg / kg / h, which is maintained until the end of surgical procedure
  Interventions: Drug: Lidocaine
- Group P (Placebo Comparator): Normal saline solution administered under the same regimen
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine — Bolus 1.5 mg/kg over 5 minutes, then an infusion of 2 mg/kg/h
  Arms: Group L
Drug: Normal saline — Sodium Chloride 0.9% infusion
  Other Names: Saline solution
  Arms: Group P

SUMMARY:
There some evidence regarding the effect of lidocaine for the prevention of nausea and vomiting in adults.

DETAILED DESCRIPTION:
The investigators want to know whether with intravenous lidocaine a adjunct for general anesthesia for children between 2 and 12 years who are undergoing tonsillectomy, with or without adenoids has the same effect.

ELIGIBILITY:
Inclusion Criteria:

* Children between 2 and 12 years
* ASA I or II
* Programmed for elective tonsillectomy with or without adenoidectomy under general anesthesia

Exclusion Criteria:

* Obesity, defined as body mass index (BMI) ≥ 95th percentile for age and sex.
* Use of antiemetic drugs during the 24 hours before surgery.
* Gastroesophageal reflux.
* History of allergy to any of the drugs used in the study.
* Down Syndrome.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Evaluating the effectiveness of intravenous lidocaine during anesthesia to decrease the numbers of events (vomiting) during the immediate postoperative period up to 24 hours postoperatively, comparing to placebo | 24 hours

SECONDARY OUTCOMES:
The prevention of the composite "nausea / or vomiting" | 24 hours
Compare frequency of vomiting by baseline risk | 24 hours
Time to first vomiting | 24 hours
Time at which discharge criteria are met Postanesthesia care unit (PACU) | 24 hours
Length of stay in PACU unit | 24 hours
PACU opioid consumption | 24 hours
Postoperative pain using Children and Infants Postoperative Pain Scale , face or Visual analogue Scale, as appropriate | 24 hours
Postoperative agitation using Pediatric Anesthesia Emergence Delirium Scale | 24 hours
Time to first emetic drug administered | 24 hours
Type and number of doses of antiemetic drug required during hospitalization | 24 hours
Total length of stay | 24 hours
Analysis of cost-effectiveness. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Fernando R Altermatt, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- División de Anestesia - Facultad de Medicina Pontificia Universidad Católica, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Derived] Echevarria GC, Altermatt FR, Paredes S, Puga V, Auad H, Veloso AM, Elgueta MF. Intra-operative lidocaine in the prevention of vomiting after elective tonsillectomy in children: A randomised controlled trial. Eur J Anaesthesiol. 2018 May;35(5):343-348. doi: 10.1097/EJA.0000000000000807. PMID 29570108